CLINICAL TRIAL: NCT06246656
Title: Hard and Soft Tissue Changes During Maxillary Expansion Using Skeletally Anchored Appliances: a Prospective, Randomized Clinical Study.
Brief Title: Evaluation of Hard and Soft Tissue Change During Maxillary Expansion Using a Computer-aided Design / Computer-aided Manufacturing Appliance.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Alexander Schwaerzler, DMD, Principal Investigator, Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1804/2022
Record Dates: First submitted 2023-03-10; First posted 2024-02-07 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Palatal Expansion Technique
Keywords: CAD/CAM; Orthodontics; Maxillary Expansion; Soft Tissue Change
MeSH Terms: interventions — Palatal Expansion Technique

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CAD/CAM milled TAD guides (Active Comparator): The position guides for orthodontic Temporary Anchorage Devices (TAD) will be produced by CAD/CAM milling.
  Interventions: Procedure: Maxillary Expansion
- 3D printed guides (Active Comparator): The position guides for orthodontic Temporary Anchorage Devices (TAD) will be produced by 3D printing technology.
  Interventions: Procedure: Maxillary Expansion

INTERVENTIONS:
Procedure: Maxillary Expansion — Palatal Expansion using a CAD/CAM appliance

SUMMARY:
* Hard tissue changes during the transversal expansion of the maxilla using a CAD/CAM expansion appliance.
* Soft tissue changes during the transversal expansion of the maxilla using a CAD/CAM expansion appliance.

Participants will undergo orthodontic treatment, including:

* Initial records (intraoral scan, CBCT (cone-beam computed tomography) scan, face scan)
* Placement of guided orthodontic TADs (Temporary Anchorage Devices)
* Skeletal expansion using CAD/CAM appliance
* Fixed multibracket appliance in the upper and lower jaw
* Intermediate and terminal documents (intraoral scan, CBCT scan, face scan)

DETAILED DESCRIPTION:
This clinical trial aims to evaluate the influence of maxillary expansion using a CAD/CAM-manufactured appliance impact on the soft and hard tissues in the midfacial region in adolescent and adult orthodontic patients.

This study aims to evaluate how this treatment changes the bony structures and soft tissues (for example, the nose) in the mid-facial region during the transversal expansion of the maxilla using a CAD/CAM expansion appliance.

The appliance consists of two anchorage elements on the first molars and two TADs. The mini-screws are placed on the palate under local anesthesia with the help of drilling templates.

CAD/CAD milled and 3D printed guides will be used for the placement of the TADs.

The study will be conducted on orthodontic patients between 12 and 26 years who will receive fixed orthodontic braces in the upper and lower jaw and show a width deficit of the upper jaw.

Intraoral, face, and computed tomography (CT) scans will be used for the investigation. An intraoral and face scanner enables a high-resolution 3D image of the teeth and face. A CBCT Scan is a three-dimensional X-ray image.

These examinations do not involve pain and are performed during regular follow-up appointments.

ELIGIBILITY:
Inclusion Criteria:

* Maxillary transverse deficit,
* Lateral crossbite

Exclusion Criteria:

* Previous orthodontic treatment,
* Craniofacial anomalies,
* Severe facial asymmetries,
* Pregnancy,
* Periodontal lesions

Ages: 12 Years to 26 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 38 (Estimated)
Dates: Start 2025-01-02 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Millimetric landmark changes of hard and soft tissue measured by the digital superimposition of CBCT Scans. | up to six months
  Comparison of midfacial landmark changes during maxillary expansion

SECONDARY OUTCOMES:
CAD/CAM milled versus 3D printed guides for orthodontic TADs compared by the millimetric and angular deviation of planned and clinical position. | up to 4 weeks
  Transfer accuracy of milled and 3D printed drilling templates

CONTACTS AND LOCATIONS:
Overall Officials: Xiaohui Rausch-Fan, Prof., Study Director — Center of Clinical Research, University Clinic of Dentistry, Medical University of Vienna; Alexander Schwärzler, DMD, Principal Investigator — Department of Orthodontics, University Clinic of Dentistry, Medical University of Vienna; Erwin Jonke, Prof., Study Chair — Department of Orthodontics, University Clinic of Dentistry, Medical University of Vienna; Sophia Panwinkler, DMD, Principal Investigator — Department of Orthodontics, University Clinic of Dentistry, Medical University of Vienna
Locations (1):
- Medical University of Vienna, Department of Orthodontics, Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No